CLINICAL TRIAL: NCT01314612
Title: An Investigation Of The Effectiveness of a Cognitive Behavioral Group Treatment Addressing Insomnia and Nightmares In Veterans With PTSD
Brief Title: Initial Study of Insomnia/Nightmare Group Treatment for Posttraumatic Stress Disorder (PTSD)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Michael E. DeBakey VA Medical Center (U.S. Federal Agency)
Responsible Party: Robert Beck, Ph.D, Postdoctoral Fellow, Michael E. DeBakey Veterans Affairs Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-28115
Record Dates: First submitted 2011-03-09; First posted 2011-03-14 (Estimated); Last update posted 2011-03-17 (Estimated); Status verified 2011-03

CONDITIONS: Insomnia; Nightmares; Posttraumatic Stress Disorder
Keywords: Insomnia; group psychotherapy; nightmares; PTSD; posttraumatic stress disorder; Veterans; cognitive-behavioral intervention
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group Intervention (Experimental): Subjects randomly assigned to this arm of the study will receive the 9-week insomnia and nightmare intervention group once per week for 90 minutes in addition to continuing treatment as usual with medical and mental health providers.
  Interventions: Behavioral: Cognitive-Behavioral Insomnia and Nightmare Group
- Treatment as Usual (No Intervention): This group is randomly assigned to receive only treatment as usual and does not receive the active intervention of the insomnia and nightmare group treatment. This treatment will be made available to these members once the study is completed

INTERVENTIONS:
Behavioral: Cognitive-Behavioral Insomnia and Nightmare Group — Group based cognitive-behavioral therapy meeting weekly for 90 minutes over the course of 9 weeks. Utilizes stimulus control, sleep scheduling, and progressive muscle relaxation to address symptoms of insomnia. Imagery rehearsal and rescripting are used to address nightmare symptoms.
  Arms: Group Intervention

SUMMARY:
Many combat Veterans suffer from posttraumatic stress disorder (PTSD), an anxiety disorder that develops after an extremely stressful event or events. PTSD is associated with problems falling asleep or staying asleep. Veterans with PTSD also commonly have nightmares from stressful experiences. These symptoms can cause problems in daily life. Behavioral treatments that do not involve taking medication have been shown to help improve problems related to sleep and nightmares. However, very few of these treatments address both sleep problems and nightmares at the same time, even though many people suffer from both problems. The purpose of this study is to examine the effectiveness of a combined treatment for sleep problems and nightmares in Veterans suffering from combat-related PTSD that is presented in a group format. The investigators hypothesize that the completion of this treatment will lead to increases in sleep quality and decreases in the frequency and severity of nightmares as measured by standard questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Must be enrolled in the Michael E. DeBakey VAMC Trauma Recovery Program and qualify for a diagnosis of combat-related PTSD related to service in Vietnam-era conflicts as measured by responses to the Clinician-Administered PTSD Scale (CAPS) and total score ≥ 50 on the Posttraumatic Stress Disorder Checklist Stressor Specific Version (PCL-S)
* Have a clinically significant sleep problem as measured by a total score > 5 on the Pittsburgh Sleep Quality Index (PSQI)
* Have a repetitive trauma-related nightmare at least once per week on average, as measured by the Nightmare Frequency Questionnaire (NFQ), and which significantly impairs sleep as measured by response ≥ 2 on question 1a of the Nightmare Effects Survey (NES)
* Be stable on current regimen of psychotropic medication (i.e., no changes to medications and/or dosages) if applicable
* Must sign consent to be audio-recorded as part of the course of the treatment

Exclusion Criteria:

* Current substance dependence
* Planned or ongoing participation in Prolonged Exposure or Cognitive Processing Therapy during treatment participation
* Organic psychosis
* Bipolar I disorder
* Epilepsy
* Currently on benzodiazepine or hypnotic medication to treat sleep
* Currently take prazosin
* Indication of undiagnosed sleep apnea defined as score ≥ .5 across items 1, 5, and 8 of the Multivariable Apnea Risk Index
* Uncontrolled sleep apnea

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-03; Primary Completion 2011-08 (Estimated); Study Completion 2011-08 (Estimated)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index, with Addendum for PTSD | baseline and 20 weeks
  Self report measure of sleep quality and degree to which sleep is affected by PTSD.
Nightmare Effects Survey | baseline and 20 weeks
  Self-report assessment of psychosocial impairment resulting from experience of nightmares
Posttraumatic Stress Disorder Checklist- Stressor Specific Version | baseline and 20 weeks
  Self-report measure of Posttraumatic Stress Disorder symptoms.

SECONDARY OUTCOMES:
Clinician Administered PTSD Scale | baseline and 10 weeks
  Structured Clinical Interview focused on symptoms of Posttraumatic Stress Disorder

CONTACTS AND LOCATIONS:
Overall Officials: Robert D Beck, Ph.D, Principal Investigator — Michael E. DeBakey VA Medical Center; Whitney L Brown, Psy.D, Principal Investigator — Michael E. DeBakey VA Medical Center
Locations (1):
- Michael E. DeBakey VA Medical Center, Houston, Texas, United States